CLINICAL TRIAL: NCT04120688
Title: 3D Autotransplantation of Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hanna Thoren MD, Professor, Chief Physcian, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T282/2019
Record Dates: First submitted 2019-09-26; First posted 2019-10-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect on surgery (Active Comparator): Duration of surgery, degree of manipulation of the transplant
  Interventions: Device: 3D generated tooth replica
- Success of transplantation (Active Comparator): Normal eruption and root development of the transplant
  Interventions: Device: 3D generated tooth replica

INTERVENTIONS:
Device: 3D generated tooth replica — 3D generated tooth replicas are compared to conventional procedure

SUMMARY:
The study aims to clarify the usefulness of 3D-printed replicas in association with autotransplantation of teeth in children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Need for tooth transplantation
* Open apex tooth available for transplantation

Exclusion Criteria:

* Facial syndrome
* Chronic facial pain
* Allergy to replica material

Ages: 9 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with healthy transplanted teeth as assessed by clinical examination at one year. | One year postoperatively
  The transplanted tooth is clinically healthy
Number of patients with healthy transplanted teeth as assessed by radiological examination at one year. | One year postoperatively
  The transplanted tooth is radiologically healthy

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Thorén, MD, Principal Investigator — University of Turku
Locations (1):
- Turku University Hospital, Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No